CLINICAL TRIAL: NCT04325906
Title: Early Prone Positioning Combined With High-Flow Nasal Cannula Versus High-Flow Nasal Cannula in COVID-19 Induced Moderate to Severe ARDS
Brief Title: Early PP With HFNC Versus HFNC in COVID-19 Induced Moderate to Severe ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19-HFNC+PP
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Prone Positioning; High Flow Nasal Cannula; Acute Respiratory Distress Syndrome; Corona Virus Infection
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- high flow nasal cannula only (Active Comparator): Receive high flow nasal cannula only
  Interventions: Device: high flow nasal cannula (HFNC)
- HFNC plus prone positioning (Experimental): Receive high flow nasal cannula plus prone positioning
  Interventions: Device: high flow nasal cannula (HFNC); Procedure: Prone positioning (PP)

INTERVENTIONS:
Device: high flow nasal cannula (HFNC) — HFNC will be initiated at 50 L/min (AIRVO2 or Optiflow, Fisher &Paykel Health care Limited., Auckland, New Zealand) with temperature set at 37 oC. Nasal cannula size will be determined by the patient's nostril size (≤ 50%). FIO2 will be adjusted to maintain SpO2 at 92% to 95%. Flow and temperature will be adjusted based on patient's comfort and clinical response.
Procedure: Prone positioning (PP) — PP will be performed before or 1 hour after meal. Before PP, all the I.V. lines and nasal cannula will be checked by clinicians. PP will be performed by patient under the supervision of clinicians. Assistance will be offered if needed. If tolerated, PP will be maintained for at least 30 minutes, until the patients feel tired to keep that position. PP will be performed twice a day for the first 3 days after the patient's enrollment. FIO2 will be adjusted to maintain SpO2 at 92-95%.
  Arms: HFNC plus prone positioning

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an emerging infectious disease that was first reported in Wuhan, China, and had subsequently spread worldwide. Twenty-nine percent of COVID-19 patients may develop ARDS. Based on the potential beneficial mechanisms of HFNC and PP, whether early use of prone positioning combined with HFNC can avoid the need for intubation in COVID-19 induced moderate to severe ARDS patients needs to be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 induced adult ARDS patients admitted to the medical ICU
* PaO2/FiO2 is less than 200mmHg or FIO2 ≥ 0.4 is required to maintain SpO2 at 88-93% on HFNC treatment

Exclusion Criteria:

1. If the patients have a consistent SpO2<80% when on evaluation with a FiO2 of 0.6, or signs of respiratory fatigue (RR > 40/min, PaCO2> 50mmHg / pH<7.30, and obvious accessory respiratory muscle use);
2. Immediate need for intubation (PaO2/FiO2< 50mmHg or SpO2/FiO2 <90, unable to protect airway or mental status change);
3. unstable hemodynamic status(SBP<90mmHg, MBP below 65 mmHg or requirement for vasopressor);
4. unable to collaborate with HFNC/PP with agitation or refuse HFNC/PP.
5. chest trauma or any contraindication for PP
6. pneumothorax
7. age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Ding L, Wang L, Ma W, He H. Efficacy and safety of early prone positioning combined with HFNC or NIV in moderate to severe ARDS: a multi-center prospective cohort study. Crit Care. 2020 Jan 30;24(1):28. doi: 10.1186/s13054-020-2738-5. PMID 32000806
- [Background] Munshi L, Del Sorbo L, Adhikari NKJ, Hodgson CL, Wunsch H, Meade MO, Uleryk E, Mancebo J, Pesenti A, Ranieri VM, Fan E. Prone Position for Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S280-S288. doi: 10.1513/AnnalsATS.201704-343OT. PMID 29068269
- [Background] Scholten EL, Beitler JR, Prisk GK, Malhotra A. Treatment of ARDS With Prone Positioning. Chest. 2017 Jan;151(1):215-224. doi: 10.1016/j.chest.2016.06.032. Epub 2016 Jul 8. PMID 27400909
- [Background] Respiratory care committee of Chinese Thoracic Society. [Expert consensus on preventing nosocomial transmission during respiratory care for critically ill patients infected by 2019 novel coronavirus pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Feb 20;17(0):E020. doi: 10.3760/cma.j.issn.1001-0939.2020.0020. Online ahead of print. Chinese. PMID 32077661
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Tavernier E, McNicholas B, Pavlov I, Roca O, Perez Y, Laffey J, Mirza S, Cosgrave D, Vines D, Frat JP, Ehrmann S, Li J. Awake prone positioning of hypoxaemic patients with COVID-19: protocol for a randomised controlled open-label superiority meta-trial. BMJ Open. 2020 Nov 11;10(11):e041520. doi: 10.1136/bmjopen-2020-041520. PMID 33177145
- [Background] Pavlov I, He H, McNicholas B, Perez Y, Tavernier E, Trump MW, Jackson JA, Zhang W, Rubin DS, Spiegel T, Hung A, Estrada MAI, Roca O, Vines DL, Cosgrave D, Mirza S, Laffey JG, Rice TW, Ehrmann S, Li J. Awake Prone Positioning in Non-Intubated Patients With Acute Hypoxemic Respiratory Failure Due to COVID-19. Respir Care. 2022 Jan;67(1):102-114. doi: 10.4187/respcare.09191. Epub 2021 Jul 7. PMID 34234032
- [Background] Li J, Pavlov I, Laffey JG, Roca O, Mirza S, Perez Y, McNicholas B, Cosgrave D, Vines D, Tavernier E, Ehrmann S. Meta-trial of awake prone positioning with nasal high flow therapy: Invitation to join a pandemic collaborative research effort. J Crit Care. 2020 Dec;60:140-142. doi: 10.1016/j.jcrc.2020.07.020. Epub 2020 Jul 24. No abstract available. PMID 32799184
- [Result] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Result] Kaur R, Vines DL, Mirza S, Elshafei A, Jackson JA, Harnois LJ, Weiss T, Scott JB, Trump MW, Mogri I, Cerda F, Alolaiwat AA, Miller AR, Klein AM, Oetting TW, Morris L, Heckart S, Capouch L, He H, Li J. Early versus late awake prone positioning in non-intubated patients with COVID-19. Crit Care. 2021 Sep 17;25(1):340. doi: 10.1186/s13054-021-03761-9. PMID 34535158

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Flow Nasal Cannula Only | HFNC Plus Prone Positioning
Started | 112 | 112
Completed | 110 | 112
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Flow Nasal Cannula Only | HFNC Plus Prone Positioning | Total
Number analyzed (Participants) | 110 | 112 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (13.3) | 62.2 (12.5) | 62.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 68 | 72 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 65 | 122
  Not Hispanic or Latino | 53 | 47 | 100
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure (Intubation or Death)
Description: the treatment failure rate of HFNC/HFNC+PP support within 28 days of study enrollment
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Nasal Cannula Only | HFNC Plus Prone Positioning
Number analyzed (Participants) | 110 | 112
Participants | 45 | 45

2. Primary Outcome: Number of Participants With Intubation
Description: intubation rate of HFNC/HFNC+PP support within 28 days of study enrollment
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Nasal Cannula Only | HFNC Plus Prone Positioning
Number analyzed (Participants) | 110 | 112
Participants | 39 | 38

3. Primary Outcome: Mortality
Description: mortality of HFNC/HFNC+PP support within 28 days of study enrollment
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Nasal Cannula Only | HFNC Plus Prone Positioning
Number analyzed (Participants) | 110 | 112
Participants | 30 | 21

4. Secondary Outcome: Number of Participants With Adverse Events
Description: adverse events include skin breakdown, vomiting, arterial or central line dislodgement, and cardiac arrest
Time Frame: 28 days of study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Nasal Cannula Only | HFNC Plus Prone Positioning
Number analyzed (Participants) | 110 | 112
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Within 28 days of study enrollment
Arm/Group | High Flow Nasal Cannula Only | HFNC Plus Prone Positioning
All-Cause Mortality (participants affected / at risk) | 30/110 | 21/112
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/112
Other Adverse Events (participants affected / at risk) | 0/110 | 2/112
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Flow Nasal Cannula Only (N=110) | HFNC Plus Prone Positioning (N=112)
Central or arterial line dislodgement (Surgical and medical procedures) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study funder (Rice foundation) had no role in study design, data analysis, the preparation or approval of the manuscript, or the decision to submit the manuscript for publication

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form: Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT04325906/Prot_ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT04325906/Prot_SAP_003.pdf